CLINICAL TRIAL: NCT02829749
Title: A European, Multicenter, Randomized Study Comparing the Effectiveness and Safety of Mitral Valve Repair With the NeoChord DS1000 Artificial Chordae Delivery System Versus Conventional Surgery in Patients With Severe Primary Mitral Regurgitation Due to Isolated Leaflet Prolapse
Brief Title: Effectiveness and Safety of Mitral Valve Repair With the NeoChord DS1000 Artificial Chordae Delivery System Versus Conventional Surgery in Patients With Severe Primary Mitral Regurgitation Due to Isolated Leaflet Prolapse
Acronym: MITRACHORD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of dynamics in the field of minimal invasive mitral repair and the development of newer devices
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL16_0115; IDRCB (Other: 2017-A01387-46)
Record Dates: First submitted 2016-07-04; First posted 2016-07-12 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Cardiovascular Diseases
Keywords: Heart Valve Diseases; Heart failure; Heart diseases; Mitral valve insufficiency
MeSH Terms: conditions — Cardiovascular Diseases; Heart Valve Diseases; Heart Failure; Heart Diseases; Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NeoChord DS1000 Artificial Chordae Delivery System (Experimental): Subjects randomized to the experimental group will undergo the NeoChord implantation
  Interventions: Device: NeoChord beating heart mitral valve implantation
- Control (Other): traditional mitral valve repair performed under cardiac arrest
  Interventions: Procedure: Control

INTERVENTIONS:
Device: NeoChord beating heart mitral valve implantation — The NeoChord DS1000 procedure is performed in five steps: (1) Device Preparation; (2) Left Ventricular Access; (3) Leaflet Capture and Verification; (4) Suture Deployment and (5) Suture Closure. The sutures are placed via a ventriculotomy 2-4 cm postero-lateral from the apex of the left ventricle via thoracotomy. The procedure is performed on a beating heart through a 2 to 3 inch right antero-lateral thoracotomy, then one to five Goretex neochordae are introduced with a transcatheter delivery system through the apex of the heart, into the left ventricle, and fixed on the free edge of the prolapsed leaflet. This is performed with transesophageal echocardiographic guidance.
  Arms: NeoChord DS1000 Artificial Chordae Delivery System
Procedure: Control — traditional mitral valve repair performed under cardiac arrest
  Arms: Control

SUMMARY:
The main objective is to assess the effectiveness and safety of the NeoChord DS1000 repair technique as compared with conventional open-heart on-pump mitral valve surgery in patients with severe primary mitral regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* Severe primary mitral regurgitation (grade 3+ or 4+)
* Class I indication for MV Surgery according to ESC/EACTS and AHA/ACC guidelines:

  1. Symptomatic patients and/or
  2. LV (Left Ventricular) dysfunction : LVESD ≥45 mm and/or 30≤ LVEF ≤60%
* Leaflet prolapse of P2 and/or A2
* Predicted coaptation length > 4 mm
* Candidates for surgical mitral valve repair according to heart team
* Patient able to sign an informed consent form
* Patient benefiting from a social insurance system or a similar system

Exclusion Criteria:

* Asymptomatic patients with preserved LV function
* Complex mechanism of MR (leaflet perforation, severe calcifications, commissural extension, etc)
* Secondary MR
* Predicted post-repair coaptation length less than 4 mm
* Atrial fibrillation
* Inflammatory or infective valve disease
* Severe LV dilation (DTD > 65 mm)
* Significant mitral annulus dilatation (D > 45 mm)
* Surgical indication of tricuspid annulus
* Contraindication to TEE (transesophageal echocardiographic ) or inadequate image quality
* Need for any other concomitant cardiac procedure
* Concurrent medical condition with a life expectancy of less than 24 months
* Patient unable to understand the purpose of the trial
* Patient < 18 years old
* Participation to another trial that would interfere with this trial
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Combined incidence of Death from any cause, redo surgery for valve dysfunction, and moderate-severe (3+) or severe (4+) mitral regurgitation | 1 year

SECONDARY OUTCOMES:
Proportion of patients with any major adverse events | 30 days
  Major adverse events defined by death all cause, Post-operative myocardial infarction, Reoperation for failed surgical repair or valve replacement, Any reoperation or intervention for adverse events (Bleeding…), stoke, renal failure, wound infection, septicemia, ventilation > 24 hours, transfusion ≥ 2 units
Overall survival | 12 months
Mitral valve reoperation free survival | 12 months
mitral regurgitation > 2+ | 12 months
Freedom from rehospitalization for heart failure | 12 months
Change in functional evaluation (NYHA) | 12 months
Change in functional evaluation (6 minute walk test ) | 12 months
Change in quality of life score | 12 months
  by using the EQ-5D questionnaire ( European Quality of Life-5 Dimensions) instrument
Number of device success | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François OBADIA, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Louis Pradel, Bron, France

IPD SHARING:
Plan to Share IPD: No